CLINICAL TRIAL: NCT00000985
Title: Treatment of Acyclovir-Resistant Mucocutaneous Herpes Simplex Infection in Patients With the Acquired Immunodeficiency Syndrome: A Randomized Multicenter Study of Foscarnet Versus Vidarabine
Brief Title: Comparison of Foscarnet Versus Vidarabine in the Treatment of Herpes Infection in Patients With AIDS Who Have Not Had Success With Acyclovir
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Model: Parallel | Purpose: Treatment
Other Study IDs: ACTG 095; 11070 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Herpes Simplex; HIV Infections
Keywords: Vidarabine; Phosphonoacetic Acid; Herpes Simplex; Foscarnet; Acyclovir; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Herpes Simplex; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Vidarabine; Acyclovir; Foscarnet

INTERVENTIONS:
Drug: Vidarabine
Drug: Acyclovir
Drug: Foscarnet sodium

SUMMARY:
To compare the safety and effectiveness of foscarnet and vidarabine treatments for AIDS patients who have herpes simplex virus infections that are resistant to standard treatment with acyclovir.

Foscarnet is a drug that inhibits viruses and has been shown to be effective against infection with Cytomegalovirus and also against infection with the Herpes simplex virus in several patients with AIDS. Vidarabine has been shown to have activity against the Herpes simplex virus in patients who do not have AIDS, but it has not been studied in patients who do have AIDS. This study compares foscarnet and vidarabine treatments for AIDS patients who have herpes simplex infection that has not responded to therapy with acyclovir in the hope that one of these two drugs will help to stop further progression of the herpes simplex infection and may have fewer side effects.

DETAILED DESCRIPTION:
Foscarnet is a drug that inhibits viruses and has been shown to be effective against infection with Cytomegalovirus and also against infection with the Herpes simplex virus in several patients with AIDS. Vidarabine has been shown to have activity against the Herpes simplex virus in patients who do not have AIDS, but it has not been studied in patients who do have AIDS. This study compares foscarnet and vidarabine treatments for AIDS patients who have herpes simplex infection that has not responded to therapy with acyclovir in the hope that one of these two drugs will help to stop further progression of the herpes simplex infection and may have fewer side effects.

Following evaluation studies, patients receive at least 10 days of intravenous (IV) therapy with acyclovir. During this therapy, patients have two serum concentration levels of acyclovir drawn to make sure there are adequate levels of medication in their blood. If skin lesions do not heal after a total of 10 days of therapy with acyclovir, lesions are swabbed for viral culture to test the susceptibility of the virus to therapy with acyclovir, foscarnet, and vidarabine. If the test confirms that the herpes lesions are resistant to acyclovir, patients may choose to participate in the next phase of the study. Following additional evaluation studies, patients are randomized to one of two groups, each of which receives 10-21 days of IV treatment with one of the two alternative medications, foscarnet or vidarabine. Foscarnet is given by IV infusion every 8 hours, and each infusion lasts 1 hour. Vidarabine is given by IV infusion once a day, and each infusion lasts 12 hours. While receiving therapy with either foscarnet or vidarabine, blood tests are done every 3 days for routine lab tests and once a week to determine foscarnet or vidarabine blood levels. Skin lesions are cultured for herpes virus every 5 days. At the end of 10 days of therapy, improvement is evaluated, and the patients can continue to receive therapy if indicated. There is a provision for cross-over treatment if patients show a poor response.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed for phase B:

* Aerosolized pentamidine prophylaxis for Pneumocystis carinii pneumonia (PCP).

Prior Medication:

Allowed for phase A:

* Ganciclovir. Patients receiving this drug at the time of study enrollment must discontinue the drug at the time of enrollment and for the duration of the study period.

Exclusion Criteria

Co-existing Condition:

For phase A, patients with pre-existing severe neurologic impairment such as seizure disorder or marked or incapacitating ataxia are excluded.

Concurrent Medication:

Excluded upon entry into phase B:

* Ganciclovir.
* Immunomodulators.
* Probenecid.
* Ciprofloxacin.
* Allopurinol.
* Zidovudine (AZT).
* Antiretrovirals.
* Other investigational agents.
* Acyclovir for another labeled indication.
* Potentially nephrotoxic agents.

Patients will be excluded from the study for the following reasons:

Phase A:

* Previous hypersensitivity reaction to foscarnet or vidarabine. Patients who have a documented history of vidarabine intolerance may be eligible for the foscarnet on the non-randomized arm of the study.

Phase B:

* Clinical response to therapy with acyclovir in phase A described as "healed" or "good."

Prior Medication:

Excluded within 14 days of study entry:

* Immunomodulators or biologic response modifiers.

Phase A:

* Excluded within 30 days of study entry:
* Foscarnet.

Phase B:

Excluded within 7 days of study entry into phase B:

* Any potentially nephrotoxic agent, except acyclovir.

Prior Treatment:

Excluded for phase A within 14 days of study entry:

* Lymphocyte replacement therapy.

Patients must demonstrate the following clinical and laboratory findings:

Phase A:

* HIV positive by federally licensed ELISA test confirmed by Western blot, p24 serum antigen, or a positive HIV culture; or a prior diagnosis of AIDS as defined by Centers for Disease Control criteria.
* Mucocutaneous herpes simplex virus (HSV) infection confirmed by viral culture persisting for a minimum of 2 weeks which is clinically resistant to therapy with acyclovir in the opinion of the patient's physician.

Phase B:

* Persistent shedding of HSV at the completion of or within 1 week after completion of phase A acyclovir therapy as confirmed by viral culture.

Documented in vitro resistance of the virus to acyclovir.

* All strains must be referred to the Diagnostic Virology Laboratories at either San Francisco General Hospital or Beth Israel Hospital, Boston, for susceptibility testing.
* Two serum acyclovir levels drawn during phase A. Results may be pending at time of entry into phase B.
* All eligibility evaluations must be performed within 7 days prior to study entry for phase A or B.

Ages: 13 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26
Dates: Study Completion 1990-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: S Safrin, Study Chair
Locations (4):
- United States (4):
  - Rush Univ. Med. Ctr. ACTG CRS, Chicago, Illinois
  - Beth Israel Deaconess - East Campus A0102 CRS, Boston, Massachusetts
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - University of Washington AIDS CRS, Seattle, Washington

REFERENCES:
- [Background] Safrin S, Crumpacker C, Chatis P, Davis R, Hafner R, Rush J, Kessler HA, Landry B, Mills J. A controlled trial comparing foscarnet with vidarabine for acyclovir-resistant mucocutaneous herpes simplex in the acquired immunodeficiency syndrome. The AIDS Clinical Trials Group. N Engl J Med. 1991 Aug 22;325(8):551-5. doi: 10.1056/NEJM199108223250805. PMID 1649971
- [Background] Safrin S, Crumpacker C, Chatis P, Davis R, Hafner R, Rush J, Kessler H, Landry B, Mills J. ACTG 095: a randomized comparison of foscarnet (FOS) vs. Vidarabine (ARA-A) for treatment of acyclovir (ACV)-resistant mucocutaneous herpes simplex virus (HSV) infection in patients with AIDS. Int Conf AIDS. 1991 Jun 16-21;7(1):44 (abstract no MB85)